CLINICAL TRIAL: NCT01401608
Title: RF Ablation of Idiopathic VT and PVCs Using Remote Magnetic Navigation
Brief Title: Stereotaxis Idiopathic Ventricular Tachycardia (VT) Study
Status: Terminated | Type: Observational
Why Stopped: Difficult to recruit eligible subjects
Sponsor: Stereotaxis (Industry)
Responsible Party: Sponsor
Other Study IDs: PM-CLIN-015
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Ventricular Tachycardia
Keywords: VT; ventricular tachycardia; ablation; magnetic navigation; robotic
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Treatment: Ablation of VT/PVCs using a magnetic RF ablation catheter
  Interventions: Device: RF Ablation

INTERVENTIONS:
Device: RF Ablation — Ablation of arrhythmogenic ventricular tissue
  Other Names: ThermoCool; Niobe; Stereotaxis

SUMMARY:
This study will assess the outcomes of using magnetic navigation to treat ventricular tachycardia (VT) or premature ventricular contractions (PVCs) that occur for unknown reasons and are not related to structural heart disease.

DETAILED DESCRIPTION:
During conventional ventricular arrhythmia ablation procedures, simply contacting the cardiac wall can significantly alter the electrocardiogram. Induction of ventricular ectopy is important in determining the focus of the arrhythmogenic tissue during an electrophysiology (EP) procedure; however, instrumentation with stiff ablation catheters can temporarily eliminate VT during the mapping portion of the procedure making it difficult to track the arrhythmia prior to ablating the tissue responsible for its genesis. The catheters used with the Stereotaxis Magnetic Navigation System (MNS) are less stiff compared to manual catheters since no pull wires are required to deflect the distal tip. Large external magnets positioned on either side of the EP procedure table create a magnetic field within the patient's chest. These large magnets (in direct relationship to the magnetic field) can be manipulated using specialized software. The physician controls the distal tip of the catheter by using the software while remotely using a catheter advancing system (QuickCAS®, Stereotaxis, Inc, St. Louis, MO) to reach the desired location within the heart. The soft catheters may provide a unique quality to the electrophysiologist who may assist by providing accurate maps without temporarily eliminating the ventricular ectopy due to excessive mechanical forces applied to the cardiac tissue. This study will assess the physician's ability to appropriately map and ablate the ventricular substrate using remote magnetic technology. All devices are approved by FDA and no off-label use of the products is mandated within the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be between 18 - 80 years of age
* Willing to provide written informed consent
* Present with ventricular ectopy of non-ischemic origin
* able to be safely exposed to a static magnetic field
* Failure of at least 1 antiarrhythmic medication

Exclusion Criteria:

* Presence of a mobile ventricular thrombus
* Unable to obtain percutaneous access to the left ventricle
* Contraindicated for short-term anticoagulation therapy
* Life expectancy less than 1 year
* Body habitus limits placement on the procedure table
* Previously failed ablation procedure for VT/PVCs

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be diagnosed with any ventricular tachycardia or symptomatic PVCs of non-ischemic origin.
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2011-03; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change in 24-hour Holter Monitor (number of extra ventricular beats) | Change from Holter Monitor Pre-procedure vs. 6-Months Post-procedure
  Use of the MNS in mapping and ablation of idiopathic VT will lead to a 75% reduction in the number of individual ventricular ectopic beats 6 months after the procedure. Extra ventricular beats will be counted using a 24-hour Holter monitor pre-procedure (obtained no more than 30 days prior to the procedure) compared to a 24-hour Holter monitor 6 months post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Raul Weiss, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States